CLINICAL TRIAL: NCT04309604
Title: IC14 for ALS Patients Expanded Access
Acronym: EAP
Status: No longer available | Type: Expanded Access
Sponsor: Implicit Bioscience (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ALS-03
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Motor Neurone Disease; Compassionate use
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: IC14 — monoclonal antibody directed against CD14

SUMMARY:
The primary objective is to provide the investigational product, IC14, at the dose of 8 mg/kg intravenously every 2 weeks for 12 weeks to 6 participants with amyotrophic lateral sclerosis (ALS). No clinical hypotheses are being tested. An extension for 6 additional doses every 2 weeks will be allowed if the drug is safe and well tolerated.A second extension for 14 doses every 2 weeks will be allowed if the drug is safe and well tolerated.

DETAILED DESCRIPTION:
Manipulation of immune-driven inflammatory responses may have therapeutic utility in amyotrophic lateral sclerosis (ALS) and recent data suggest that ALS may respond to peripheral intervention by expanding Tregs in mice and humans. The approach with IC14 builds on this hypothesis by targeting CD14 as a master regulator of the immune response of peripheral cell populations, which in turn determines the activation status and phenotype of peripheral T cells that enter the central nervous system (CNS) and drive further microglia activation .Binding and blocking membrane CD14 (mCD14) on peripheral immune cell populations with IC14 may thus be a relevant therapeutic target in ALS.

IC14 has been safe, well tolerated and had no serious adverse events related to study drug.

This is a protocol for 12 weeks of the investigational medication IC14 for 6 participants. An extension for 6 additional doses every 2 weeks will be done if the drug is safe and well tolerated. Up to 20 subjects may be screened in order to identify eligible subjects that meet all inclusion and exclusion criteria.

At the screening visit, the Principal Investigator will review the study procedures and consent form with the participant. After obtaining informed consent, the participant will receive IC14 8 mg/kg intravenously every two weeks (± 7 days) for 6 doses (12 weeks). An extension for 6 additional doses every 2 weeks will be allowed if the drug is safe and well tolerated. A second extension for 14 additional doses every 2 weeks will be allowed if the drug is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any program-specific procedures.
2. Familial or sporadic ALS defined as clinically possible, probable, or definite by Awaji-Shima Consensus Recommendations or other standard guidance.
3. Adequate hematologic, renal, and liver function as defined by the patient's physician.
4. Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods:

   1. Sexual abstinence (inactivity) for 1 month prior to screening through study completion; or
   2. Intrauterine device (IUD) in place for at least 3 months prior to study through study completion; or
   3. Stable hormonal contraception for at least 3 months prior to study through study completion; or
   4. Surgical sterilization (vasectomy) of male partner at least 6 months prior to study.
5. To be considered of non-childbearing potential, females should be surgically sterilized (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be post-menopausal and at least 3 years since last menses.
6. Males with female partners of childbearing potential must use contraception through study completion.

Exclusion Criteria:

1. Dependence on invasive mechanical ventilation, defined as being unable to lay supine without it, unable to sleep without it, or continuous daytime use; presence of tracheostomy at screening;
2. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other opportunistic infections; or major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of baseline.
3. Immunized with live-attenuated vaccines within 30 days before dosing. Participants must agree to forego live-attenuated vaccines throughout the program, including 12 weeks after the last dose of IC14.
4. History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
5. Pregnancy or breastfeeding.
6. Presence of any of the following clinical conditions:

   * History of one or more of the following: cardiac insufficiency (New York Heart Association III/IV), uncontrolled cardiac arrhythmias, unstable ischemic heart disease, or uncontrolled hypertension (systolic blood pressure > 170 mmHg or diastolic blood pressure > 110 mmHg).
   * History of venous thromboembolic disease within 6 months, myocardial infarction, or cerebrovascular accident.
   * Unstable pulmonary, renal, hepatic, endocrine or hematologic disease.
   * Autoimmune disease, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis.
   * Evidence of active malignant disease, malignancies diagnosed within the previous 5 years, or breast cancer diagnosed within the previous 5 years (except skin cancers other than melanoma).
   * History of human immunodeficiency virus infection or other immunodeficiency illness.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gelevski D, Addy G, Rohrer M, Cohen C, Roderick A, Winter A, Carey J, Scalia J, Yerton M, Weber H, Doyle M, Parikh N, Kane G, Ellrodt A, Burke K, D'Agostino D, Sinani E, Yu H, Sherman A, Agosti J, Redlich G, Charmley P, Crowe D, Appleby M, Ziegelaar B, Hanus K, Li Z, Babu S, Nicholson K, Luppino S, Berry J, Baecher-Allan C, Paganoni S, Cudkowicz M. Safety and activity of anti-CD14 antibody IC14 (atibuclimab) in ALS: Experience with expanded access protocol. Muscle Nerve. 2023 May;67(5):354-362. doi: 10.1002/mus.27775. Epub 2022 Dec 30. PMID 36533976